CLINICAL TRIAL: NCT03142971
Title: Focused Extracorporeal Shock Wave Therapy for Greater Trochanteric Pain Syndrome With Gluteal Tendinopathy: a Randomized Controlled Trial
Brief Title: Shock Wave Therapy for Lateral Hip Pain, Caused by Tendon Pathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Ettore Carlis, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20130001077
Record Dates: First submitted 2017-04-28; First posted 2017-05-08 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Tendinopathy
Keywords: Shock waves; Greater trochanteric pain syndrome
MeSH Terms: conditions — Tendinopathy | interventions — Extracorporeal Shockwave Therapy; Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Intervention:f-ESWT (focused shock wave therapy) (Experimental): In the study-group, a device powered by a piezoelectric generator (PIEZOSON 100PLUS, Richard Wolf) was used . At the beginning of each treatment session, the enthesis of the gluteal tendons at the greater trochanter (at the anterior half of its lateral facet) was targeted through a non-inline sonographic focusing, using a linear probe (7.5-12 MHz) connected to an ultrasound scanner (ESAOTE MYLAB FIVE, Genova and Florence, Italy). All patients received 1800 pulses (frequency=4Hz) of an energy flux density of 0.15 mJ/mm2 once a week for three consecutive weeks. At the first treatment session, the energy flux density was gradually increased from 0.05 to 0.15 mJ/mm2 during the first 500 pulses.
  Interventions: Procedure: focused shock wave therapy
- Intervention:UST (ultrasound therapy) (Active Comparator): In the control-group, we used a mono-frequency device (ROLAND, RT-20 series, frequency=1MHz). We treated an area of 5cm2, softly moving the US-probe around the most painful point of the greater trochanter at the clinical palpation. UST was supplied in a continuous modality, with an intensity of 1.5 W/cm2, for ten consecutive daily sessions of ten minutes each.
  Interventions: Procedure: ultrasound therapy

INTERVENTIONS:
Procedure: focused shock wave therapy
  Arms: Intervention:f-ESWT (focused shock wave therapy)
Procedure: ultrasound therapy
  Arms: Intervention:UST (ultrasound therapy)

SUMMARY:
The aim of this randomized controlled study is to investigate if focal shock wave is an effective treatment, with respect to hip pain and lower limb function, in a population affected by greater trochanteric pain syndrome with gluteal tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* duration of lateral hip pain of six weeks or longer,
* normal passive hip range of movement (ROM),
* sonographic evidence of gluteal tendinopathy at their insertional site at the greater trochanter

Exclusion Criteria:

* general contraindication to extracorporeal shock wave therapy (pacemaker, pregnancy, bleeding disorders or anticoagulant drug usage, cancer in the focal area),
* history of rheumatologic disease,
* previous fractures or surgery in the affected limb,
* full thickness tear of the gluteal tendons,
* osteoarthritis of the hip (with ROM limitation),
* clinical signs of lumbar radiculopathy,
* corticosteroid injections or other conservative therapies (except pharmacological pain treatments) since the onset of the current pain episode.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-05-04 (Actual); Study Completion 2016-05-04 (Actual)

PRIMARY OUTCOMES:
p-NRS | Baseline, at two months, at six months
  Change from baseline p-NRS (pain-on-movement numeric rating scale) at 2 months and at 6 months.
LEFS score | Baseline, at two months, at six months
  Change from baseline LEFS (Lower extremity functional scale) total score at 2 months and at 6 months